CLINICAL TRIAL: NCT00167531
Title: The Efficacy of Treadmill Training in Establishing Walking After Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sydney (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02/06/09
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2009-10-02 (Estimated); Status verified 2006-09

CONDITIONS: Stroke
Keywords: Stroke; health outcomes; physiotherapy; rehabilitation; treadmill
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treadmill walking (Experimental): 30 minutes per day of treadmill walking with body weight support and assistance from one therapist
  Interventions: Behavioral: treadmill walking with partial weight support
- Overground walking (Active Comparator): 30 minutes per day of overground walking with assistance from one therapist
  Interventions: Behavioral: assisted overground walking

INTERVENTIONS:
Behavioral: treadmill walking with partial weight support
  Arms: Treadmill walking
Behavioral: assisted overground walking — 30 minutes per day of overground walking with the assistance of one therapist
  Arms: Overground walking

SUMMARY:
Being able to walk is a major determinant of whether a patient returns home after stroke or lives in residential care. For the family, the loss of the stroke sufferer from everyday life is a catastrophic event. For the community, the costs of being unable to walk after stroke are exorbitant, involving a lifetime of residential care. Therefore, an increase in the proportion of stroke patients who regain walking ability will be a significant advance.

This trial will determine, in patients early after stroke who are unable to walk, whether training walking using a treadmill with partial weight support via an overhead harness will be more effective than current intervention in (i) establishing more independent walking, reducing the time taken to achieve independent walking, and improving the quality of independent walking, and (ii) improving walking capacity and participation 6 months later.

DETAILED DESCRIPTION:
Only half of the stroke patients unable to walk who are admitted to inpatient rehabilitation in Australia learn to walk again. Treadmill training with partial weight support is a relatively new intervention that is designed to train walking. However, a Cochrane Systematic Review (Moseley et al 2003) concludes that there is as yet no definitive answer about whether this intervention helps more non-ambulatory patients learn to walk compared to assisted overground walking.

Participants will be 130 stroke patients who are unable to walk independently early after stroke. They will be recruited and randomly allocated to a control group or an experimental group.

The control group will undertake routine assisted overground walking training while the experimental group will undertake treadmill walking with partial weight support via an overhead harness. Duration and frequency of intervention and the amount of assistance from therapists will be standardised across groups.

ELIGIBILITY:
Inclusion Criteria:

* First stroke
* Within 28 days post stroke
* Aged between 50 and 85 years of age
* Unilateral hemiplegia/hemiparesis and
* Score for Item 5 of the Motor Assessment Scale for Stroke < 2

Exclusion Criteria:

* Any barriers to taking part in a physical rehabilitation program
* Insufficient cognition/language
* Unstable cardiac status
* Neuro-surgery
* Any pre-morbid history of orthopaedic conditions or any other problems that would preclude patient from relearning to walk.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2002-08; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Proportion of participants walking independently (defined for the purposes of this study as'being able to walk 15 m continuously across flat ground without any aids'). | Within 6 months

SECONDARY OUTCOMES:
Quality of walking: measured by quantifying parameters such as speed, affected and intact step length, step width, and cadence during 10 m walk test. | Within 6 months
Walking capacity at six months measured by 10 m and 6 minute walk tests. Walking participation measured using the Adelaide Activity Profile. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Louise Ada, PhD, Principal Investigator — University of Sydney; Catherine Dean, PhD, Principal Investigator — University of Sydney; Meg Morris, PhD, Principal Investigator — University of Melbourne; Judy Simpson, PhD, Principal Investigator — University of Sydney
Locations (5):
- Australia (5):
  - The Prince Henry and Prince of Wales Hospitals, Sydney, New South Wales
  - Royal Rehabilitation Centre Sydney, Sydney, New South Wales
  - Blacktown / Mt Druitt Hospital, Sydney, New South Wales
  - St George Hospital, Sydney, New South Wales
  - Kingston Centre, Melbourne, Victoria

REFERENCES:
- [Background] Ada L, Dean CM, Hall JM, Bampton J, Crompton S. A treadmill and overground walking program improves walking in persons residing in the community after stroke: a placebo-controlled, randomized trial. Arch Phys Med Rehabil. 2003 Oct;84(10):1486-91. doi: 10.1016/s0003-9993(03)00349-6. PMID 14586916
- [Derived] Dean CM, Ada L, Bampton J, Morris ME, Katrak PH, Potts S. Treadmill walking with body weight support in subacute non-ambulatory stroke improves walking capacity more than overground walking: a randomised trial. J Physiother. 2010;56(2):97-103. doi: 10.1016/s1836-9553(10)70039-4. PMID 20482476
- [Derived] Ada L, Dean CM, Morris ME, Simpson JM, Katrak P. Randomized trial of treadmill walking with body weight support to establish walking in subacute stroke: the MOBILISE trial. Stroke. 2010 Jun;41(6):1237-42. doi: 10.1161/STROKEAHA.109.569483. Epub 2010 Apr 22. PMID 20413741
- [Derived] Ada L, Dean CM, Morris ME. Supported treadmill training to establish walking in non-ambulatory patients early after stroke. BMC Neurol. 2007 Sep 6;7:29. doi: 10.1186/1471-2377-7-29. PMID 17803825